CLINICAL TRIAL: NCT03109548
Title: Pre-treatment Factors for the Development of Chronic Pain in Low Back Pain Patients
Status: Completed | Type: Observational
Sponsor: Aalborg University (Other)
Collaborators: Research Unit for General Practice in Aalborg (Other)
Responsible Party: Principal Investigator, Kristian Kjær Petersen, assistant professor, Aalborg University
Other Study IDs: N-20160086
Record Dates: First submitted 2017-03-31; First posted 2017-04-12 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Standard care initiated by the general practitioner — Patients are treated based on their symptoms and the research group does not interfere with this.

SUMMARY:
The purpose of the project is to associate pre-treatment pain sensitivity level, levels of pain catastrophizing and levels of The Subgroups for Targeted Treatment (STarT) Back Screening Tool in patients with acute low back pain and patients' progression after 12 weeks of treatment by general practitioners.

ELIGIBILITY:
Inclusion Criteria:

* Patients with low back pain, who have a mobile phone.

Exclusion Criteria:

* Pregnancy
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Alcohol addiction
* Lack of ability to cooperate
* Surgery to the spine

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The subjects will be recruited through general practitioners in The North Denmark Region. When a patient with low back pain reports to his/her general practitioner, the doctor will present the project to the patient, and in case the patient shows interest, the doctor asks him/her to contact the contact person of the study. Thus, the recruitment does not take place through advertisements, but through the normal patient flow in the general practice.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2018-11-06 (Actual)

PRIMARY OUTCOMES:
Roland Morris Disability Questionnaire, RMDQ | 12 weeks follow-up
  Change in the Roland-Morris Questionnaire (RMDQ) is one of the most widely used questionnaires for back pain. The RMDQ is a self-administered disability questionnaire consisting of 24 questions. The questions are related specifically to physical functions likely to be affected by low back pain. Each item is qualified with the phrase "because of my back pain" to distinguish back pain disability from disability due to other causes. When completing the RMDQ, the respondents are asked to tick a statement if it applies to them on that particular day.

SECONDARY OUTCOMES:
The StarT Back Screening Tool | Baseline, 12 weeks follow-up
  The The StarT Back Screening Tool (SBST) is a nine-item patient self-reporting questionnaire validated for triage of nonspecific low back pain patients in primary care.
The Pain Catastrophizing Scale | Baseline, 12 weeks follow-up
  The Pain Catastrophizing Scale (PCS) consists of 13 items focusing on thoughts and feelings in connection with pain.
Predicting the Inception of Chronic Pain | Baseline, 12 weeks follow-up
  The Predicting the Inception of Chronic Pain (PICKUP) questionnaire focuses on pain ("How much low back pain have you had during the past week?", 1 = none, 2 = very mild, 3 = mild, 4 = moderate, 5 = severe, 6 = very severe), radiating pain to the legs ("Do you have leg pain?" 0 = no, 1 = yes), compensability ("Is your back pain compensable, e.g. through worker's compensation or third party insurance?" 0 = no, 1 = yes), depression ("How much have you been bothered by feeling depressed in the past week (0-10 scale)?" 0 = not at all, 10 = extremely) and the subject's overall evaluation of the risk of chronic pain ("In your view, how large is the risk that your current pain may become persistent (0-10 scale)?" 0 = none, 10 = extreme).
Basic information | Baseline, 12 weeks follow-up
  A general questionnaire has been created for this study to gain a basic understanding of the patient's current pain, demographic information and use of medication
Assessment of the Pain Area | Baseline, 12 weeks follow-up
  Patients will be asked to draw the pain area of their low back pain on a body map.
Cuff Algometry | Baseline, 12 weeks follow-up
  Cuff algometry will be applied to assess pressure pain thresholds, temporal summation of pain and conditioned pain modulation.
Handheld Algometry | Baseline, 12 weeks follow-up
  Handheld algometry will be applied to assess pressure pain thresholds.

CONTACTS AND LOCATIONS:
Overall Officials: Martin B Jensen, MD, PhD, Principal Investigator — Research Unit for General Practice in Aalborg, Department of Clinical Medicine, Aalborg University, Aalborg, Denmark
Locations (1):
- Lægerne Sløjfen, Aalborg, Aalborg East, Denmark

IPD SHARING:
Plan to Share IPD: No